CLINICAL TRIAL: NCT02532309
Title: A 2-year, Open-label, Randomized Study to Evaluate the Efficacy of Rosuvastatin Dosing Adjustment by LDL-C Level Compared to That of 5mg Maintenance Dose in Chinese Patients With Carotid Atherosclerotic Plaques
Brief Title: A Study to Evaluate the Efficacy and Safety of Rosuvastatin in the Treatment of the Carotid Atherosclerotic Plaques
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wei Liu (Other)
Collaborators: University of Washington (Other); AstraZeneca (Industry); Beijing Clinstech-med consulting Co., Ltd (Other)
Responsible Party: Sponsor-Investigator, Wei Liu, Attending Doctor, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJFH-20150203-CAP
Record Dates: First submitted 2015-07-30; First posted 2015-08-25 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Carotid Atherosclerosis
Keywords: Rosuvastatin; Carotid Atherosclerosis plaque; Crestor; Rosuvastatin calcium
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rosuvastatin dose adjustment (Experimental)
  Interventions: Drug: Rosuvastatin (5mg，10mg，20mg)
- Rosuvastatin fixed dose (Experimental)
  Interventions: Drug: Rosuvastatin 5mg

INTERVENTIONS:
Drug: Rosuvastatin (5mg，10mg，20mg) — Rosuvastatin dose adjusted by LDL-c level( If LDL-C>1.1mmol/L and <1.8mmol/L, administrated as 5mg/day.If LDL-C ≥1.8mmol/L, adjusted every 4 weeks as 5mg，10mg，20mg.
  Arms: Rosuvastatin dose adjustment
Drug: Rosuvastatin 5mg — Rosuvastatin 5mg/day
  Arms: Rosuvastatin fixed dose

SUMMARY:
This is a 2-year, open-label, randomized study to evaluate the efficacy of Rosuvastatin dosing adjustment by LDL-C level compared to that of 5mg maintenance dose in chinese patients with Carotid Atherosclerosis.

DETAILED DESCRIPTION:
This will be a 2-year, randomized, open-label, prospective, parallel-group study. It only be held in China-Japan Friendship Hospital. Subjects with Carotid Atherosclerosis Plaques who meet all inclusion and none of the exclusion criteria will be randomized in a 1:1 ratio to receive treatment of rosuvastatin (5 mg, 10mg, 20mg) dosing adjustment by LDL-c level or fixed dose 5 mg. The study will consist of two phases: the Screening/Baseline period（-1to week 0）and the Follow-up period(0 to month 24). The follow-up period will comprise seven visits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or legal guardian can understand and sign the written informed consent form;
* LDL-C≥100mg/dl（2.6mmol/l）.
* Subjects with carotid atherosclerotic non-calcified plaques determined by color Doppler ultrasound on carotid. ( Plaque defined as limited intima media thickness≥1.5mm, according to the procedure of vascular ultrasound examination in 2009 Chinese Journal of Ultrasonography )
* Subjects had not been treated with statins, or one had been treated with antihyperlipidemics no more than 3 months within 12 months prior to screening.

Exclusion Criteria:

* Subjects known to be allergic to the study medication, or any components .
* Uncontrolled hypothyroidism defined as the systolic blood pressure(SBP) >180 mmHg or the diastolic blood pressure(DBP) >100 mmHg.
* Concomitant with severe or frequent arrhythmia, such as Atrial Fibrillation, second or third degree Atrioventricular Block, Sick sinus Syndrome etc.
* Alanine aminotransaminase (ALT) and /or Aspartate aminotransferase (AST) >1.5×ULN (upper limit of normal).
* Subjects with myopathies，or the value of Creatine kinase >1.5×ULN (upper limit of normal).
* Concomitant with chronic wasting diseases, whose life span was anticipated no longer than 2 years.
* Pregnant or nursing woman, and subjects with a Pregnant plan during this study.
* Cognitive impairment, which may affect obtaining informed consent and participating in the study procedures.
* Unwilling to receive treatment or examinations outlined in protocol.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Total Carotid Plaque Area | Up to 24 months
  A comparison of the change in total Carotid Plaques area from the two treatment groups examined by color Doppler ultrasound.
Total Carotid Plaque Area | Up to 12 months
  Reversal of total Carotid Atherosclerosis Plaques in the two rosuvastatin dose group at 12 months.

SECONDARY OUTCOMES:
Total Carotid Plaque Area | Baseline to 12 months and 24 months
  Changes from baseline in total Carotid Atherosclerosis Plaques (TPA) from the two rosuvastatin treatment groups from baseline at 12 months and 24 months.
Carotid Intima-Media Thickness(IMT) | Baseline to 12 months and 24 months
  Changes of Carotid Intima-Media Thickness (IMT) in the two rosuvastatin treatment groups from baseline to 12 months and to 24 months.
The level of Blood lipid | baseline and 1, 2, 3, 6, 12, 18, 24 months post-dose
  Changes from baseline in the level of Blood lipid from the two rosuvastatin treatment groups.
Low density lipoprotein-cholesterol (LDL-c) | Baseline to 12 months and 24 months
  Analysis of the corrlation between LDL-c and TPA from the two rosuvastatin treatment groups.
Carotid Intima-Media Thickness(IMT) | Up to 24 months
  Analysis of the corrlation between IMT and TPA in each treatment group.
Incidence of Adverse Events | Baseline to 24 months
  The categories and incidences of Adverse Events from the two treatment groups.
Incidences of Major Adverse Cardiovascular and Cerebrovascular Events（MACCE） | Baseline to 24 months
  Incidences of Major adverse cardiovascular and cerebrovascular events from the two rosuvastatin treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China